CLINICAL TRIAL: NCT00980798
Title: Randomized, Double-blind, Placebo-controlled, Parallel-group Trial to Investigate the Analgesic Effect of OROS Hydromorphone Hydrochloride in Comparison With Placebo in Subjects With Moderate to Severe Pain Induced by Osteoarthritis of the Hip or the Knee
Brief Title: Placebo-controlled Trial With OROS Hydromorphone Hydrochloride to Treat Patients With Moderate to Severe Pain Induced by Osteoarthritis of the Hip or the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR012601; HOP Trial
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Results first posted 2010-09-06 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Pain; Osteoarthritis, Hip; Osteoarthritis, Knee
Keywords: Osteoarthritis; Strong pain killer; Strong opioid; Low starting dose; Fewer side effects; Physical functioning; Pain control; Quality of life; Sleep quality
MeSH Terms: conditions — Pain; Osteoarthritis, Hip; Osteoarthritis, Knee; Osteoarthritis; Agnosia; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): OROS hydromorphone HCl 4 to 32 mg taken orally once daily for 16 weeks
  Interventions: Drug: OROS hydromorphone HCl
- 002 (Placebo Comparator): Placebo placebo tablet once daily for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OROS hydromorphone HCl — 4 to 32 mg taken orally once daily for 16 weeks
  Arms: 001
Drug: Placebo — placebo tablet once daily for 16 weeks
  Arms: 002

SUMMARY:
This clinical trial tests the pain relieving effectiveness of OROS hydromorphone, a once-daily formulation of a strong opioid against placebo in patients, who are suffering from pain due to osteoarthritis of the hip or the knee and who previously did not receive any strong opioids.The clinical trial tests the effect of the treatment on symptoms of pain, stiffness and physical function. The effect of the treatment on parameters on health related quality of life as well as quality of sleep will be measured.

DETAILED DESCRIPTION:
In this clinical trial subjects are enrolled, who are suffering from pain due to osteoarthritis of the hip or the knee that is not sufficiently controlled with either a non steroidal anti-inflammatory drug (NSAID) or paracetamol or a weak opioid. This clinical trial tests the pain relieving effectiveness of OROS hydromorphone, a once-daily formulation of a strong opioid against placebo in patients, who previously did not receive any strong opioids. The drug class of opioid analgesics can broadly be classified into strong and weak. Weak opioids (for example tramadol, codeine, dihydrocodeine and tilidine) are useful for mild to moderate pain and the strong opioids (for example morphine, fentanyl and hydromorphone) are useful for moderate to severe pain of different origin. OROS hydromorphone is an opioid, which is available in a prolonged-release tablet in different dosage strengths. The primary aim of the study is to test the efficacy of OROS hydromorphone against placebo at an individual dose sufficient to control the pain and to establish the usefulness of a new low-dose formulation of OROS hydromorphone (4 mg hydromorphone per tablet) for initiating the treatment and for dose titration. The clinical trial tests the effect of the treatment on symptoms of pain, stiffness and physical function. The effect of the treatment on parameters on health related quality of life as well as quality of sleep will be measured. The safety of the treatment will be recorded by measuring blood pressure, heart rate, and respiratory rate.This clinical trial is a placebo-controlled trial, meaning that one group of patients will receive the drug to be tested (OROS hydromorphone) while the control group receives an optically identical tablet with no active ingredient, a so-called placebo. A total number of 270 patients will be enrolled in this clinical trial and assigned to one of two treatment arms at an equal ratio (i.e. 135 patients per treatment). Patients will be randomly assigned to one of the two treatment arms, like flipping a coin to decide which treatment they will receive. Neither the patient nor the doctor will know to which of the two treatment arms the patient is assigned to and neither the patient nor the doctor can influence the assignment to the treatment arm. During the whole treatment period paracetamol will be allowed to be taken as needed in case of pain. Medical history and physical exam will be conducted during the screening visit, followed in 1 week by the baseline visit where after completing several questionnaires assessing pain, physical functioning quality of life and sleep quality, the patient will be assigned to one of two treatment groups. After starting the study treatment the patient will visit the doctor 7 times: at week 1, 2, 3, 4, 8, 12, 16 and at a follow-up visit after the end of the treatment period at week 16. At week 16 questionnaires will again be completed and the results will be compared to the baseline findings. 4, 8, 12, 16, 24 or 32 mg of OROS hydromorphone tablets or matching placebo tablets taken for 16 weeks. All tablets are taken by mouth at the same time each day in the morning. Tablets have to be swallowed whole without chewing or crushing. After completion of the treatment duration (or at early withdrawal), the study medication is gradually tapered down over a maximum of 6 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented Osteoarthritis of the hip or knee
* Chronic pain for more than 3 months treated with daily analgesic for the last month
* Moderate to severe OA pain of the target joint, which cannot be adequately treated with non-steroidal anti-inflamatory drugs or paracetamol
* Moderate to severe pain by means of a mean weekly score of >= 5 in the Brief Pain Invetory item 5 'pain on average'

Exclusion Criteria:

* Regular treatment with an opioid in the 4 weeks before screening visit (infrequent use of tramadol, codeine, tilidine, or dihydrocodeine for no more than 10 days in the 4 weeks before the screening visit is acceptable, however, treatment must be stopped at screening visit)
* Diagnosis of major depression
* Treatment for epilepsy
* Corticosteroid injection within the last 3 months
* Major surgery in the 3 months before the start of the study
* Women who are pregnant or breast-feeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (12):
- Czechia (5):
  - Klatovy
  - Olomouc
  - Pelhøimov
  - Prague
  - Roudnice nad Labem
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Iași
- Slovakia (3):
  - Bratislava
  - Hlohovec
  - Piešťany
- London, United Kingdom

REFERENCES:
- See also: Placebo-controlled trial with OROS hydromorphone hydrochloride to treat patients with moderate to severe pain induced by osteoarthritis of the hip or the knee. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=48&filename=CR012601_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject attended the first study visit on 05 October 2007, and the last subject completed the last study visit on 24 November 2008.
Groups:
- Placebo: Placebo daily for 16 weeks
Period: Overall Study
Arm/Group | Placebo | OROS Hydromorphone HCl
Started | 149 | 139
Completed | 116 | 84
Not Completed | 33 | 55
Not completed — Adverse Event | 7 | 36
Not completed — Lack of Efficacy | 16 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 8 | 11
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | OROS Hydromorphone HCl | Total
Number analyzed (Participants) | 149 | 139 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (10.37) | 65.1 (9.96) | 65 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 107 | 208
  Male | 48 | 32 | 80

OUTCOME MEASURES:

1. Primary Outcome: Analgesic Effect as Assessed by Brief Pain Inventory (BPI) Item 5 Score (Pain on Average)
Description: The analgesic effect was assessed by the BPI item 5 "pain on average" using a 0 to 10 numeric rating scale, with 0 being "no pain" and 10 being "pain as bad as you can imagine".
Time Frame: At each study visit from screening to week 16
Population: The primary population for the efficacy analyses was the intention to treat (ITT) population: all randomised patients who received at least one dose of study drug excluding patients who had no post-baseline efficacy data. This population included patients who discontinued early owing to lack of efficacy or other reasons.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | OROS Hydromorphone HCl
Number analyzed (Participants) | 143 | 132
units on a scale
  Screening | 6.4 (0.94) | 6.4 (1.05)
  Baseline (Visit 1) | 6.5 (0.94) | 6.6 (1.04)
  Visit 2 | 5.2 (1.43) | 5.0 (1.63)
  Visit 3 | 4.8 (1.66) | 4.6 (1.66)
  Visit 4 | 4.3 (1.72) | 4.0 (1.85)
  Visit 5 | 3.9 (1.9) | 3.9 (2.02)
  Visit 6 | 3.7 (1.97) | 3.5 (1.88)
  Visit 7 | 3.6 (1.99) | 3.4 (1.96)
  Visit 8 | 4.0 (2.3) | 4.1 (2.2)
  Visit 9 | 4.2 (2.27) | 4.4 (2.23)
Statistical Analysis 1: Comparison: Placebo vs OROS Hydromorphone HCl; The F test for treatment tested the null hypothesis of no treatment difference. Assuming that 3 baseline measures and 7 post baseline measures were collected 81 patients were required per group to detect a difference of 1 point in the BPI measure with 90% power at a significance level of 5%. To allow for a drop-out rate of approximately 40%, the study planned to recruit 135 patients per group (i.e. 270 in total); Test type: Superiority or Other; p = 0.1212, Mixed-model regression analysis — No adjustment for multiple comparisons necessary, as only 1 primary hypothesis was tested. Threshold for statistical significance was 0.05; The difference above is presented as the difference OROS hydromorphone HCl minus placebo, so negative scores favour OROS hydromorphone HCl; Mean Difference (Net) = -0.2365, 95% CI 2-sided [-0.5357 to 0.0627] — The analysis was adjusted for baseline BPI item 5 score, time on study, and whether the primary affected joint was the hip or knee

2. Secondary Outcome: The Number of Patients Discontinuing From the Trial Due to the Occurrence of an Adverse Event
Description: The number of patients dropping out of the study owing to adverse events will be presented for each treatment group.
Time Frame: At each study visit from baseline until week 16
Population: Safety population: All randomised patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | OROS Hydromorphone HCl
Number analyzed (Participants) | 149 | 139
participants | 7 | 36

ADVERSE EVENTS:
Time Frame: Adverse were collected from signing of informed consent until the end of the study (week 16 or later after complete tapering off of study medication)
Arm/Group | Placebo | OROS Hydromorphone HCl
Serious Adverse Events (participants affected / at risk) | 7/149 | 4/139
Other Adverse Events (participants affected / at risk) | 50/149 | 106/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=149) | OROS Hydromorphone HCl (N=139)
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Cardioversion (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=149) | OROS Hydromorphone HCl (N=139)
Constipation (Gastrointestinal disorders) | 10 | 63
Nausea (Gastrointestinal disorders) | 10 | 41
Vomiting (Gastrointestinal disorders) | 2 | 15
Dry mouth (Gastrointestinal disorders) | 7 | 11
Somnolence (Nervous system disorders) | 22 | 45
Dizziness (Nervous system disorders) | 5 | 15
Headache (Nervous system disorders) | 4 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 10
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 7
Vertigo (Ear and labyrinth disorders) | 4 | 10
Anorexia (Metabolism and nutrition disorders) | 1 | 8

LIMITATIONS AND CAVEATS:
Concomitant and rescue medication were permitted in the study. This may be why the results in the placebo arm so closely resemble those in the treatment arm. Patients were also less severely impacted by the underlying disease than in other studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days